CLINICAL TRIAL: NCT02588300
Title: Evaluation of the Upper Airway Collapse in Patients With Obstructive Sleep Apnea Syndrome by Drug Induced Sleep Endoscopy According to the Munich Sleep Video Protocol
Brief Title: Upper Airway Collapse in Patients With Obstructive Sleep Apnea Syndrome by Drug Induced Sleep Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5782/13
Record Dates: First submitted 2015-10-25; First posted 2015-10-27 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug induced sleep endoscopy (Experimental): Patients upper airway is assessed by drug induced sleep endoscopy
  Interventions: Procedure: Drug induced sleep endoscopy

INTERVENTIONS:
Procedure: Drug induced sleep endoscopy — Titration of propofol using a target controlled Infusion pump and description of the upper airway according to the VOTE classification

SUMMARY:
This is a prospective, interventional cohort study of drug-induced sleep endoscopy (DISE). The goal is to evaluate the upper airway in a cohort of patients with obstructive sleep apnea hypopnea syndrome (OSAHS) diagnosed in a prior polysomnography.

This study correlates the sedation level measured by entropy during DISE using propofol via a TCI pump with the local obstruction patterns of the upper airway according to the VOTE classification.

As OSAHS is a widespread disease and the DISE procedure has become a common tool for diagnosis and evaluation of further treatment, a growing number of research articles deal with this topic. These articles are available through pubmed.

ELIGIBILITY:
Inclusion Criteria:

* documented sleep apnea Syndrome with an AHI > 5 diagnosed by polysomnography

Exclusion Criteria:

* active infection
* performed oral, head or neck surgery, pregnancy,
* ASA classification III or higher,
* chronic use of alcohol, sedatives or illicit drugs and chronic
* obstructive pulmonary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
collapse of the upper airway according to the VOTE classification | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Edenharter, MD, Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Klinik für Anaesthesiologie, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Heiser C, Fthenakis P, Hapfelmeier A, Berger S, Hofauer B, Hohenhorst W, Kochs EF, Wagner KJ, Edenharter GM. Drug-induced sleep endoscopy with target-controlled infusion using propofol and monitored depth of sedation to determine treatment strategies in obstructive sleep apnea. Sleep Breath. 2017 Sep;21(3):737-744. doi: 10.1007/s11325-017-1491-8. Epub 2017 Mar 31. PMID 28364198